CLINICAL TRIAL: NCT01174420
Title: A Prospective Randomized Comparative Study of the Safety and Effectiveness of Ologen Collagen Matrix Versus Mitomycin-C in Trabeculectomy
Brief Title: Comparative Study of Ologen Collagen Matrix Versus Mitomycin-C in Trabeculectomy: A Study in Germany
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aeon Astron Europe B.V. (Industry)
Responsible Party: Thomas Dietlein, Department of Ophthalmology, University of Cologne, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAE-CT-DEU-2009-01
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Open-angle Glaucoma
Keywords: ologen; Mitomycin-C; Collagen Matrix; trabeculectomy; glaucoma; filtering surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ologen Collagen Matrix (Experimental)
  Interventions: Device: Use of ologen Collagen Matrix in trabeculectomy
- Mitomycin-C (MMC) (Active Comparator)
  Interventions: Drug: Use of Mitomycin-C in trabeculectomy

INTERVENTIONS:
Device: Use of ologen Collagen Matrix in trabeculectomy — After trabeculectomy, place ologen Collagen Matrix on the top of the scleral flap under the conjunctiva before suturing
  Arms: ologen Collagen Matrix
Drug: Use of Mitomycin-C in trabeculectomy — After creating a scleral flap, a sponge with Mitomycin-C (0.02%) is applied on the scleral surface for 3 minutes. Afterwards, Mitomycin-C was rinsed out with balanced salt solution.
  Arms: Mitomycin-C (MMC)

SUMMARY:
The aim of this prospective randomized study is to investigate the efficacy and safety of trabeculectomy with ologen Collagen Matrix versus trabeculectomy using mitomycin C (MMC) in patients with medically uncontrolled open angle glaucoma.

DETAILED DESCRIPTION:
ologen® Collagen Matrix (CM) is an artificial extracellular matrix (ECM) specifically configured to support repair in connective and epithelial ocular tissue. The device is constructed so as to minimize random growth of fibroblasts and instead to allow them to grow through the pores in the matrix. ologen® CM is a biodegradable scaffold matrix, inducing a regenerative non-scarring wound healing process without using anti-fibrotic agents. For application in glaucoma filtration surgery, ologen® CM is designed to prevent scar formation (subconjunctival and scleral flap scarring is the major risk factor for failure of trabeculectomy). After implanting the ologen® CM on top of the scleral flap in the subconjunctival space, a functional bleb can be created.

The aim of the present study is to determine the effectiveness of the ologen® CM and reduce wound scarring, thereby increasing success of trabeculectomy without side effects of MMC. A means of producing better success rate and reduced complications is the purpose of ologen® Collagen Matrix for the aid of glaucoma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Uncontrolled open-angle glaucoma
* Subject is willing to sign informed consent
* Subject is able and willing to complete post-operative follow-up requirements

Exclusion Criteria:

* Inflammatory eye diseases
* Angle-closure glaucoma
* Secondary glaucoma with anatomical malformations of the eye
* Subjects having single functional eye
* Previous conjunctival surgery
* Known allergic reactions to ingredients of ologen Collagen Matrix
* Excessive myopia (axial length (AL)> 27 mm or more than -10 diopters)
* Previous vitrectomy eye surgery
* Subjects do not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) reduction | 6 months

SECONDARY OUTCOMES:
Incidence of complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietlein, MD, Principal Investigator — Department of Ophthalmology, University of Cologne, Germany
Locations (1):
- The University Hospital of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740